CLINICAL TRIAL: NCT02014519
Title: Seroprevalence of Bordetella Pertussis in Adults in Hungary
Brief Title: A Study to Determine the Seroprevalence of Bordetella Pertussis in Adults in Hungary
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 116804
Record Dates: First submitted 2013-12-12; First posted 2013-12-18 (Estimated); Results first posted 2018-12-17 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Pertussis; Pertussis Vaccines
Keywords: Adults; Hungary; Bordetella pertussis; Seroprevalence; Pertussis antibodies
MeSH Terms: conditions — Whooping Cough | interventions — Blood Specimen Collection; Data Collection

ARMS (1):
- Study Group (Other): Subjects, male and female, aged 18 years and above who had agreed to collection of blood sample.
  Interventions: Procedure: Blood sampling; Other: Data collection

INTERVENTIONS:
Procedure: Blood sampling — A blood sample (2.5 mL) will be collected from all subjects
Other: Data collection — Active questioning

SUMMARY:
The purpose of this study is to perform an epidemiological survey of the adult population in Hungary to calculate the seroprevalence of pertussis.

DETAILED DESCRIPTION:
The protocol posting was amended to correct the detailed title. Since a sample of blood will be collected from all subjects (outside of routine hospital procedure), the study does not meet GSK's definition of an observational study and hence the term "observational" was deleted from the detailed title.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* Written informed consent will be obtained from subjects prior to performing any study procedures.
* Males or females ≥ 18 years of age at the time of enrollment.
* Agreeing to collection of a blood sample for the study.

Exclusion Criteria:

• Confirmed or suspected immunological disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2014-04-24 (Actual); Primary Completion 2015-04-22 (Actual); Study Completion 2015-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Hungary (4):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Kecskemét
  - GSK Investigational Site, Zirc

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/SearchAllPostings.aspx?searchparam=116804

REFERENCES:
- [Background] Torzsa P, Devadiga R, Tafalla M. Seroprevalence of Bordetella pertussis antibodies in adults in Hungary: results of an epidemiological cross-sectional study. BMC Infect Dis. 2017 Apr 4;17(1):242. doi: 10.1186/s12879-017-2356-2. PMID 28376739

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Group
Started | 2000
Completed | 2000
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Group
Number analyzed (Participants) | 2000
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (17.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1213
  Male | 787
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Seropositive Subjects in Terms of Anti-pertussis Toxin (Anti-PT) Concentrations
Description: Seropositivity was defined as anti-PT IgG levels above the sensitivity limit of the assay (> 0.3 Optical Density (OD) units)
Time Frame: At the time of enrollment of each subject (Day 0)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort included all evaluable subjects for whom valid laboratory test results for anti-pertussis toxin antibodies were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 1999
Participants | 295

2. Primary Outcome: Number of Subjects With Anti-PT IgG Levels Strongly Indicative of Current/Recent Infection
Description: The cut-off value for anti-PT IgG levels strongly indicative of current/recent infection was greater than or equal to (≥) 1.5 OD units
Time Frame: At the time of enrollment of each subject (Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 1999
Participants | 2

3. Primary Outcome: Number of Subjects With Anti-PT IgG Levels Indicative of Current/Recent Infection
Description: The cut-off value for anti-PT IgG levels indicative of current/recent infection was greater than or equal to (≥) 1.0 OD units.
Time Frame: At the time of enrollment of each subject (Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 1999
Participants | 22

4. Primary Outcome: Number of Seronegative Subjects in Terms of Anti-PT Concentrations
Description: Seronegativity was defined as anti-PT IgG levels under the sensitivity limit of the assay (≤ 0.3 OD units)
Time Frame: At the time of enrollment of each subject (Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 1999
Participants | 1704

5. Secondary Outcome: Number of Seropositive Subjects in Terms of Anti-PT Concentrations (by Age)
Description: Seropositivity was defined as anti-PT IgG levels above the sensitivity limit of the assay (> 0.3 OD units).
Time Frame: At the time of enrollment of each subject (Day 0).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- 18-29 Years Group: Subjects, male and female, aged 18-29 years at the time of enrollment, who had agreed to collection of blood sample.
- 30-44 Years Group: Subjects, male and female, aged 30-44 years at the time of enrollment, who had agreed to collection of blood sample.
- 45-59 Years Group: Subjects, male and female, aged 45-59 years at the time of enrollment, who had agreed to collection of blood sample.
- ≥ 60 Years Group: Subjects, male and female, aged 60 years and above at the time of enrollment, who had agreed to collection of blood sample.
Arm/Group | 18-29 Years Group | 30-44 Years Group | 45-59 Years Group | ≥ 60 Years Group
Number analyzed (Participants) | 408 | 541 | 509 | 541
Participants | 67 | 67 | 56 | 105

6. Secondary Outcome: Number of Subjects With Anti-PT IgG Levels Strongly Indicative of Current/Recent Infection (by Age)
Description: as for outcome 2
Time Frame: At the time of enrollment of each subject (Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 18-29 Years Group | 30-44 Years Group | 45-59 Years Group | ≥ 60 Years Group
Number analyzed (Participants) | 408 | 541 | 509 | 541
Participants | 0 | 1 | 1 | 0

7. Secondary Outcome: Number of Subjects With Anti-PT IgG Levels Indicative of Current/Recent Infection (by Age)
Description: as for outcome 3
Time Frame: At the time of enrollment of each subject (Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 18-29 Years Group | 30-44 Years Group | 45-59 Years Group | ≥ 60 Years Group
Number analyzed (Participants) | 408 | 541 | 509 | 541
Participants | 2 | 5 | 4 | 11

8. Secondary Outcome: Number of Seronegative Subjects in Terms of Anti-PT Concentrations (by Age)
Description: Seronegativity was defined as anti-PT IgG levels under the sensitivity limit of the assay (≤ 0.3 OD units)
Time Frame: At the time of enrollment of each subject (Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 18-29 Years Group | 30-44 Years Group | 45-59 Years Group | ≥ 60 Years Group
Number analyzed (Participants) | 408 | 541 | 509 | 541
Participants | 341 | 474 | 453 | 436

9. Secondary Outcome: Number of Seropositive Subjects in Terms of Anti-PT Concentrations (by Gender)
Description: Seropositivity was defined as anti-PT IgG levels above the sensitivity limit of the assay (> 0.3 OD units)
Time Frame: At the time of enrollment of each subject (Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Female Group: Female subjects aged 18 years and above who had agreed to collection of blood sample.
- Male Group: Male subjects aged 18 years and above who had agreed to collection of blood sample.
Arm/Group | Female Group | Male Group
Number analyzed (Participants) | 1212 | 787
Participants | 160 | 135

10. Secondary Outcome: Number of Subjects With Anti-PT IgG Levels Strongly Indicative of Current/Recent Infection (by Gender)
Description: as for outcome 2
Time Frame: At the time of enrollment of each subject (Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Female Group | Male Group
Number analyzed (Participants) | 1212 | 787
Participants | 0 | 2

11. Secondary Outcome: Number of Subjects With Anti-PT IgG Levels Indicative of Current/Recent Infection (by Gender)
Description: as for outcome 3
Time Frame: At the time of enrollment of each subject (Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Female Group | Male Group
Number analyzed (Participants) | 1212 | 787
Participants | 10 | 12

12. Secondary Outcome: Number of Seronegative Subjects in Terms of Anti-PT Concentrations (by Gender)
Description: Seronegativity was defined as anti-PT IgG levels under the sensitivity limit of the assay (≤ 0.3 OD units)
Time Frame: At the time of enrollment of each subject (Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Female Group | Male Group
Number analyzed (Participants) | 1212 | 787
Participants | 1052 | 652

13. Secondary Outcome: Number of Subjects With Anti-PT IgG Levels Not Indicative of Current/Recent Infection (by Gender)
Description: The cut-off value for anti-PT IgG levels not indicative of current/recent infection was smaller than (<) 1.0 OD units.
Time Frame: At the time of enrollment of each subject (Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Male Group | Female Group
Number analyzed (Participants) | 787 | 1212
Participants | 775 | 1202

14. Secondary Outcome: Number of Seropositive Subjects in Terms of Anti-PT Concentrations (by Recent History of Long-lasting Cough)
Description: Seropositivity was defined as anti-PT IgG levels above the sensitivity limit of the assay (> 0.3 OD units). A long-lasting cough was defined as any cough that lasted for more than (≥) 3 weeks in the previous 12 months.
Time Frame: At the time of enrollment of each subject (Day 0)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort included all evaluable subjects for whom valid laboratory test results for anti-pertussis toxin antibodies were available and who provided information on recent history of long-lasting cough.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 1795
Participants
  Without long-lasting cough: number analyzed (Participants) | 1568
  Without long-lasting cough | 240
  With long-lasting cough: number analyzed (Participants) | 227
  With long-lasting cough | 30

15. Secondary Outcome: Number of Seronegative Subjects in Terms of Anti-PT Concentrations (by Recent History of Long-lasting Cough)
Description: Seronegativity was defined as anti-PT IgG levels under the sensitivity limit of the assay (≤ 0.3 OD units). A long-lasting cough was defined as any cough that lasted for more than (≥) 3 weeks in the previous 12 months.
Time Frame: At the time of enrollment of each subject (Day 0)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 1795
Participants
  Without long-lasting cough: number analyzed (Participants) | 1568
  Without long-lasting cough | 1328
  With long-lasting cough: number analyzed (Participants) | 227
  With long-lasting cough | 197

16. Secondary Outcome: Number of Subjects With Anti-PT IgG Levels Indicative of Current/Recent Infection (by Recent History of Long-lasting Cough)
Description: The cut-off value for anti-PT IgG levels indicative of current/recent infection was greater than or equal to (≥) 1.0 OD units. A long-lasting cough was defined as any cough that lasted for more than (≥) 3 weeks in the previous 12 months.
Time Frame: At the time of enrollment of each subject (Day 0)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 1795
Participants
  Without long-lasting cough: number analyzed (Participants) | 1568
  Without long-lasting cough | 17
  With long-lasting cough: number analyzed (Participants) | 227
  With long-lasting cough | 4

17. Secondary Outcome: Number of Subjects With Anti-PT IgG Levels Not Indicative of Current/Recent Infection (by Recent History of Long-lasting Cough)
Description: The cut-off value for anti-PT IgG levels not indicative of current/recent infection was smaller than (<) 1.0 OD units. A long-lasting cough was defined as any cough that lasted for more than (≥) 3 weeks in the previous 12 months.
Time Frame: At the time of enrollment of each subject (Day 0)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 1795
Participants
  Without long-lasting cough: number analyzed (Participants) | 1568
  Without long-lasting cough | 1551
  With long-lasting cough: number analyzed (Participants) | 227
  With long-lasting cough | 223

18. Secondary Outcome: Number of Seropositive Subjects in Terms of Anti-PT Concentrations (by Smoking Status)
Description: Seropositivity was defined as anti-PT IgG levels above the sensitivity limit of the assay (> 0.3 OD units)
Time Frame: At the time of enrollment of each subject (Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 1999
Participants
  Never Smoker: number analyzed (Participants) | 1079
  Never Smoker | 136
  Former Smoker: number analyzed (Participants) | 482
  Former Smoker | 86
  Current Smoker: number analyzed (Participants) | 438
  Current Smoker | 73

19. Secondary Outcome: Number of Seronegative Subjects in Terms of Anti-PT Concentrations (by Smoking Status)
Description: Seronegativity was defined as anti-PT IgG levels under the sensitivity limit of the assay (≤ 0.3 OD units)
Time Frame: At the time of enrollment of each subject (Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 1999
Participants
  Never Smoker: number analyzed (Participants) | 1079
  Never Smoker | 943
  Former Smoker: number analyzed (Participants) | 482
  Former Smoker | 396
  Current Smoker: number analyzed (Participants) | 438
  Current Smoker | 365

20. Secondary Outcome: Number of Subjects With Anti-PT IgG Levels Indicative of Current/Recent Infection (by Smoking Status)
Description: as for outcome 3
Time Frame: At the time of enrollment of each subject (Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 1999
Participants
  Never Smoker: number analyzed (Participants) | 1079
  Never Smoker | 4
  Former Smoker: number analyzed (Participants) | 482
  Former Smoker | 8
  Current Smoker: number analyzed (Participants) | 438
  Current Smoker | 10

21. Secondary Outcome: Number of Subjects With Anti-PT IgG Levels Not Indicative of Current/Recent Infection (by Smoking Status)
Description: The cut-off value for anti-PT IgG levels not indicative of current/recent infection was smaller than (<) 1.0 OD units.
Time Frame: At the time of enrollment of each subject (Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 1999
Participants
  Never Smoker: number analyzed (Participants) | 1079
  Never Smoker | 1075
  Former Smoker: number analyzed (Participants) | 482
  Former Smoker | 474
  Current Smoker: number analyzed (Participants) | 438
  Current Smoker | 428

22. Secondary Outcome: Number of Seropositive Subjects in Terms of Anti-PT Concentrations (by History of Pertussis)
Description: Seropositivity was defined as anti-PT IgG levels above the sensitivity limit of the assay (> 0.3 OD units)
Time Frame: At the time of enrollment of each subject (Day 0)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort included all evaluable subjects for whom valid laboratory test results for anti-pertussis toxin antibodies were available and who provided information on history of pertussis.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 1566
Participants
  Without history of Pertussis: number analyzed (Participants) | 1478
  Without history of Pertussis | 212
  With history of Pertussis: number analyzed (Participants) | 88
  With history of Pertussis | 15

23. Secondary Outcome: Number of Seronegative Subjects in Terms of Anti-PT Concentrations (by History of Pertussis)
Description: Seronegativity was defined as anti-PT IgG levels under the sensitivity limit of the assay (≤ 0.3 OD units)
Time Frame: At the time of enrollment of each subject (Day 0)
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 1566
Participants
  Without history of Pertussis: number analyzed (Participants) | 1478
  Without history of Pertussis | 1266
  With history of Pertussis: number analyzed (Participants) | 88
  With history of Pertussis | 73

24. Secondary Outcome: Number of Subjects With Anti-PT IgG Levels Indicative of Current/Recent Infection (by History of Pertussis)
Description: as for outcome 3
Time Frame: At the time of enrollment of each subject (Day 0)
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 1566
Participants
  Without history of Pertussis: number analyzed (Participants) | 1478
  Without history of Pertussis | 18
  With history of Pertussis: number analyzed (Participants) | 88
  With history of Pertussis | 1

25. Secondary Outcome: Number of Subjects With Anti-PT IgG Levels Not Indicative of Current/Recent Infection (by History of Pertussis)
Description: The cut-off value for anti-PT IgG levels not indicative of current/recent infection was smaller than (<) 1.0 OD units.
Time Frame: At the time of enrollment of each subject (Day 0)
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 1566
Participants
  Without history of Pertussis: number analyzed (Participants) | 1478
  Without history of Pertussis | 1460
  With history of Pertussis: number analyzed (Participants) | 88
  With history of Pertussis | 87

26. Secondary Outcome: Number of Seropositive Subjects in Terms of Anti-PT Concentrations (by History of Vaccination Against Pertussis)
Description: Seropositivity was defined as anti-PT IgG levels above the sensitivity limit of the assay (> 0.3 OD units)
Time Frame: At the time of enrollment of each subject (Day 0)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort included all evaluable subjects for whom valid laboratory test results for anti-pertussis toxin antibodies were available and who provided information on history of vaccination against pertussis.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 1163
Participants
  Without history of vaccination against Pertussis: number analyzed (Participants) | 281
  Without history of vaccination against Pertussis | 38
  With history of vaccination against Pertussis: number analyzed (Participants) | 882
  With history of vaccination against Pertussis | 127

27. Secondary Outcome: Number of Seronegative Subjects in Terms of Anti-PT Concentrations (by History of Vaccination Against Pertussis)
Description: Seronegativity was defined as anti-PT IgG levels under the sensitivity limit of the assay (≤ 0.3 OD units)
Time Frame: At the time of enrollment of each subject (Day 0)
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 1163
Participants
  Without history of vaccination against Pertussis: number analyzed (Participants) | 281
  Without history of vaccination against Pertussis | 243
  With history of vaccination against Pertussis: number analyzed (Participants) | 882
  With history of vaccination against Pertussis | 755

28. Secondary Outcome: Number of Subjects With Anti-PT IgG Levels Indicative of Current/Recent Infection (by History of Vaccination Against Pertussis)
Description: as for outcome 3
Time Frame: At the time of enrollment of each subject (Day 0)
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 1163
Participants
  Without history of vaccination against Pertussis: number analyzed (Participants) | 281
  Without history of vaccination against Pertussis | 2
  With history of vaccination against Pertussis: number analyzed (Participants) | 882
  With history of vaccination against Pertussis | 7

29. Secondary Outcome: Number of Subjects With Anti-PT IgG Levels Not Indicative of Current/Recent Infection (by History of Vaccination Against Pertussis)
Description: The cut-off value for anti-PT IgG levels indicative of current/recent infection was smaller than (<) 1.0 OD units.
Time Frame: At the time of enrollment of each subject (Day 0)
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 1163
Participants
  Without history of vaccination against Pertussis: number analyzed (Participants) | 281
  Without history of vaccination against Pertussis | 279
  With history of vaccination against Pertussis: number analyzed (Participants) | 882
  With history of vaccination against Pertussis | 875

30. Secondary Outcome: Number of Seropositive Subjects in Terms of Anti-PT Concentrations (by Medication)
Description: Seropositivity was defined as anti-PT IgG levels above the sensitivity limit of the assay (> 0.3 OD units). Medication included any antibiotics and/or other medication (i.e. any cough medicines) for lower respiratory tract infections, Pertussis infections or suspected Pertussis infections in the previous 12 months.
Time Frame: At the time of enrollment of each subject (Day 0)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort included all evaluable subjects for whom valid laboratory test results for anti-pertussis toxin antibodies were available and who provided information on their medication history.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 1962
Participants
  Without history of medication: number analyzed (Participants) | 1721
  Without history of medication | 248
  With history of medication: number analyzed (Participants) | 241
  With history of medication | 39

31. Secondary Outcome: Number of Seronegative Subjects in Terms of Anti-PT Concentrations (by Medication)
Description: Seronegativity was defined as anti-PT IgG levels under the sensitivity limit of the assay (≤ 0.3 OD units). Medication included any antibiotics and/or other medication (i.e. any cough medicines) for lower respiratory tract infections, Pertussis infections or suspected Pertussis infections in the previous 12 months.
Time Frame: At the time of enrollment of each subject (Day 0)
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 1962
Participants
  Without history of medication: number analyzed (Participants) | 1721
  Without history of medication | 1473
  With history of medication: number analyzed (Participants) | 241
  With history of medication | 202

32. Secondary Outcome: Number of Subjects With Anti-PT IgG Levels Indicative of Current/Recent Infection (by Medication)
Description: The cut-off value for anti-PT IgG levels indicative of current/recent infection was greater than or equal to (≥) 1.0 OD units. Medication included any antibiotics and/or other medication (i.e. any cough medicines) for lower respiratory tract infections, Pertussis infections or suspected Pertussis infections in the previous 12 months.
Time Frame: At the time of enrollment of each subject (Day 0)
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 1962
Participants
  Without history of medication: number analyzed (Participants) | 1721
  Without history of medication | 18
  With history of medication: number analyzed (Participants) | 241
  With history of medication | 3

33. Secondary Outcome: Number of Subjects With Anti-PT IgG Levels Not Indicative of Current/Recent Infection (by Medication)
Description: The cut-off value for anti-PT IgG levels indicative of current/recent infection was smaller than (<) 1.0 OD units. Medication included any antibiotics and/or other medication (i.e. any cough medicines) for lower respiratory tract infections, Pertussis infections or suspected Pertussis infections in the previous 12 months.
Time Frame: At the time of enrollment of each subject (Day 0)
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 1962
Participants
  Without Medication: number analyzed (Participants) | 1721
  Without Medication | 1703
  With Medication: number analyzed (Participants) | 241
  With Medication | 238

34. Secondary Outcome: Number of Seropositive Subjects in Terms of Anti-PT Concentrations (by Hospitalization)
Description: Seropositivity was defined as anti-PT IgG levels above the sensitivity limit of the assay (> 0.3 OD units). History of hospitalization was defined as hospitalization due to respiratory infections in the previous 12 months.
Time Frame: At the time of enrollment of each subject (Day 0)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort included all evaluable subjects for whom valid laboratory test results for anti-pertussis toxin antibodies were available and who provided information on their hospitalization history.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 1994
Participants
  Without history of hospitalization: number analyzed (Participants) | 1984
  Without history of hospitalization | 290
  With history of hospitalization: number analyzed (Participants) | 10
  With history of hospitalization | 4

35. Secondary Outcome: Number of Seronegative Subjects in Terms of Anti-PT Concentrations (by Hospitalization)
Description: Seronegativity was defined as anti-PT IgG levels under the sensitivity limit of the assay (≤ 0.3 OD units). History of hospitalization was defined as hospitalization due to respiratory infections in the previous 12 months.
Time Frame: At the time of enrollment of each subject (Day 0)
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 1994
Participants
  Without history of hospitalization: number analyzed (Participants) | 1984
  Without history of hospitalization | 1694
  With history of hospitalization: number analyzed (Participants) | 10
  With history of hospitalization | 6

36. Secondary Outcome: Number of Subjects With Anti-PT IgG Levels Indicative of Current/Recent Infection (by Hospitalization)
Description: The cut-off value for anti-PT IgG levels indicative of current/recent infection was greater than or equal to (≥) 1.0 OD units. History of hospitalization was defined as hospitalization due to respiratory infections in the previous 12 months.
Time Frame: At the time of enrollment of each subject (Day 0)
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 1994
Participants
  Without history of hospitalization: number analyzed (Participants) | 1984
  Without history of hospitalization | 22
  With history of hospitalization: number analyzed (Participants) | 10
  With history of hospitalization | 0

37. Secondary Outcome: Number of Subjects With Anti-PT IgG Levels Not Indicative of Current/Recent Infection (by Hospitalization)
Description: The cut-off value for anti-PT IgG levels not indicative of current/recent infection was smaller than (<) 1.0 OD units. History of hospitalization was defined as hospitalization due to respiratory infections in the previous 12 months.
Time Frame: At the time of enrollment of each subject (Day 0)
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 1994
Participants
  Without history of hospitalization: number analyzed (Participants) | 1984
  Without history of hospitalization | 1962
  With history of hospitalization: number analyzed (Participants) | 10
  With history of hospitalization | 10

ADVERSE EVENTS:
Time Frame: Day 0 (all study procedures were performed and completed at the first and only visit in this study)
Description: Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | Study Group
All-Cause Mortality (participants affected / at risk) | 0/2000
Serious Adverse Events (participants affected / at risk) | 0/2000
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.